CLINICAL TRIAL: NCT02312505
Title: Estimation of Cardiac Output by a New Semi-invasive Monitoring System: Accuracy and Limitations
Brief Title: Comparison of a New Semi-invasive Monitoring System With Transpulmonary Thermodilution in Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Ole Broch, MD, Ole Broch M.D., University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AZ 162/10; AZ 162/10 (Registry Identifier: Ethical Commitee of the CAU)
Record Dates: First submitted 2012-12-03; First posted 2014-12-09 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Cardiac Output, High
Keywords: cardiac output monitoring; semi-invasive pulse contour analysis; transpulmonary thermodilution
MeSH Terms: conditions — Cardiac Output, High

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- COPFX (Other): cardiac output by PulsioFlex® Monitoring system (COPFX)
  Interventions: Device: COPFX

INTERVENTIONS:
Device: COPFX — cardiac Output by semi-invasive pulse contour analysis

SUMMARY:
The aim of the study is to investigate the accuracy of a new semi-invasive cardiac output monitoring system in patients undergoing elective cardiac surgery. The investigators hypothesize that the semi-invasive device may be affected by mean arterial pressure and systemic vascular resistance.

DETAILED DESCRIPTION:
A recently introduced semi-invasive monitoring system consists of an algorithm that provides beat-to-beat measurement of CI by analysis of the arterial blood pressure tracing. By using the autocalibration mode this software calculates the individual aortic compliance and systemic vascular resistance by taking patient data like age, height, weight and gender into account. After estimation of beat-to-beat stroke volume, a subsequent multiplication by the heart rate delivers pulse contour cardiac index. Furthermore, this device offers the opportunity for external calibration by a reference technique, e.g. pulmonary or transpulmonary thermodilution.

The aim of the present study was to investigate the accuracy and trending ability of autocalibrated semi-invasive CI by a new arterial waveform analysis compared with transpulmonary thermodilution before and after cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective coronary artery bypass grafting Personal declaration of consent to the study

Exclusion Criteria:

Patients <18 years of age A left ventricular ejection fraction ≤0.5 Emergency procedures Patients with haemodynamic instability requiring continuous pharmacologic support Patients with intracardiac shunts Severe aortic-, tricuspid- or mitral stenosis or insufficiency Mechanical circulatory support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
cardiac output by pulse contour Analysis compared with transpulmonary thermodilution | participants will be followed for the start and the end of operation, on the average of 4 hours
  plotting cardiac output by a questionnaire, Statistics: correlation coefficients, Bland-Altman Analysis, trending ability by four Quadrant plots

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Bein, Professor, Study Director — University Schleswig-Holstein, Campus Kiel, Germany
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Broch O, Carbonell J, Ferrando C, Metzner M, Carstens A, Albrecht M, Gruenewald M, Hocker J, Soro M, Steinfath M, Renner J, Bein B. Accuracy of an autocalibrated pulse contour analysis in cardiac surgery patients: a bi-center clinical trial. BMC Anesthesiol. 2015 Nov 26;15:171. doi: 10.1186/s12871-015-0153-2. PMID 26612072